CLINICAL TRIAL: NCT03557047
Title: Preliminary Study on the Pathogenesis of Acute Kidney Injury After Cardiac Surgery
Brief Title: Perioperative Mechanism of Acute Kidney Injury in Cardiovascular Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Anhui Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PJ2018-03-10
Record Dates: First submitted 2018-06-03; First posted 2018-06-14 (Actual); Last update posted 2018-07-03 (Actual); Status verified 2018-03

CONDITIONS: Pathogenesis; Acute Kidney Injury; Cardiac Surgery
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Continuous observation of acute renal injury after cardiac surgery, at the same time retention of blood samples, to test indicators，and to select the research route from the clinical actual test results .

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing selective cardiac surgery, aged between 18 and 80.

Exclusion Criteria:

* Normal range of creatinine before operation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Perioperative data were collected, including cardiopulmonary bypass time，aortic cross-clamping time, operative time, extubation time, ICU time and hospital stay.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-03-08 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Incidence of acute renal injury after cardiac surgery | 48 hours
  The standard of acute renal injury is based on the KDIGO

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China